CLINICAL TRIAL: NCT03307681
Title: Effect of White Potatoes on Glycemic Response, Satiety and Food Intake in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Nick Bellissimo, Associate Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: REB2017-330 II
Record Dates: First submitted 2017-09-29; First posted 2017-10-12 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-03

CONDITIONS: Healthy
Keywords: White potatoes; Children; Satiety; Glycaemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- White bread (Experimental): Matched for energy content and available carbohydrate content of potato treatments
  Interventions: Other: White bread
- Baked potato with skin (Experimental): Baked russet potato
  Interventions: Other: Baked potato with skin
- Mashed potato served hot (Experimental): Mashed potatoes prepared from frozen, matched for available carbohydrate content of baked potato
  Interventions: Other: Mashed potato served hot
- Fried French fries (Experimental): Matched for available carbohydrate content of baked potato
  Interventions: Other: Fried French fries
- Meal skipping (Experimental): No food given
  Interventions: Other: Meal skipping

INTERVENTIONS:
Other: White bread — Toasted, with canola oil added to match for fat content of French fries (13.9 grams), as well as being matched for energy (280 kilocalories) and available carbohydrate content (33 grams) of potato treatments.
  Arms: White bread
Other: Baked potato with skin — Baked russet potato with canola oil added once baked to match for fat content of French fries, and also matched for the salt content of white bread (280 milligrams).
  Arms: Baked potato with skin
Other: Mashed potato served hot — Mashed potatoes prepared from frozen, with canola oil added to match for fat content of French fries, as well as being matched for energy and available carbohydrate content of the baked potato.
  Arms: Mashed potato served hot
Other: Fried French fries — Prepared from frozen, matched for energy and available carbohydrate content of baked potato and salt content of white bread.
  Arms: Fried French fries
Other: Meal skipping — No food given
  Arms: Meal skipping

SUMMARY:
The purpose of the present study is to explore the influence of cooking methods on post-prandial glycaemia and its impact on satiety in children.

DETAILED DESCRIPTION:
Each of the 5 study sessions will be at least 7 days apart. Either meal skipping, or one of three treatments of white potatoes (a) baked (with skin), (b) mashed, (c) fried French fries, or white bread, prepared on the day of testing, will be served to healthy children (9-14 years). Participants will consume the equivalent to 1 medium sized potato (~280 kcal) or an equivalent amount of calories from white bread. Glycemic response, insulin, incretin hormones (glucagon-like peptide-1 (GLP-1), glucose-dependent insulinotropic peptide (GIP)), dipeptidyl peptidase 4 (DPP4), and cholecystokinin (CCK) will be measured for 2 h (0, 15, 30, 45, 60, 90 and 120 min) following meal consumption, as well as mood and subjective appetite. An ad libitum test meal will be provided at 120 min to assess food intake suppression.

ELIGIBILITY:
Inclusion Criteria:

* be between 9 and 14 years of age
* be healthy, and have been born at term
* be a native English speaker
* not be taking any medications
* not have allergies to potatoes, rice, or beans.
* normal body weight (between the 5th and 85th BMI percentile for age and gender)

Exclusion Criteria:

* anyone with food sensitivities or allergies to potatoes or potato-products,
* smokers
* diabetic or overweight/obese individuals.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2020-06-21 (Actual); Study Completion 2020-06-21 (Actual)

PRIMARY OUTCOMES:
Ad libitum food intake (lunch, at 120 minutes) | at 120 minutes post morning meal consumption
  Food intake will be determined by weighing the meal before and after serving. The net weight of the test meal will be converted to calories
Change from baseline glycemic response | 15, 30, 45, 60, 90, and 120 minutes after meal consumption
  Blood glucose (mmol/L). Blood glucose will be measured in whole blood using YSI 2300 STAT PLUS (YSI Incorporated, Yellow Springs, OH)
Change from baseline insulin | 15, 30, 45, 60, 90, and 120 minutes after meal consumption
  Blood insulin (pmol/L). Insulin concentration in serum will be determined in duplicate via enzyme-linked immunosorbent assay kits (ELISA; Millipore, Billerica, Massachusetts).

SECONDARY OUTCOMES:
Change from baseline subjective appetite | 15, 30, 45, 60, 90, and 120 minutes after meal consumption
  Measured using visual analogue scale (mm). Each VAS is a 100 mm line where they will place a pencil mark to describe their feelings.
Change from baseline mood | 15, 30, 45, 60, 90, and 120 minutes after meal consumption
  Measured using visual analogue scale (mm). Each VAS is a 100 mm line where they will place a pencil mark to describe their feelings.
Change from baseline cholecystokinin (CCK) | 15, 30, 45, 60, 90, and 120 minutes after meal consumption
  Blood CCK (pmol/L). CCK concentration in serum will be determined in duplicate via enzyme-linked immunosorbent assay kits (ELISA; Millipore, Billerica, Massachusetts).
Change from baseline dipeptidyl peptidase 4 (DPP4) | 15, 30, 45, 60, 90, and 120 minutes after meal consumption
  Blood DPP4 (ng/mL). DPP4 concentration in serum will be determined in duplicate via enzyme-linked immunosorbent assay kits (ELISA; Millipore, Billerica, Massachusetts).
Change from baseline glucose-dependent insulinotropic peptide (GIP) | 15, 30, 45, 60, 90, and 120 minutes after meal consumption
  Blood GIP (pmol/L). GIP concentration in serum will be determined in duplicate via enzyme-linked immunosorbent assay kits (ELISA; Millipore, Billerica, Massachusetts).
Change from baseline glucagon-like peptide-1 (GLP-1) | 15, 30, 45, 60, 90, and 120 minutes after meal consumption
  Blood GLP-1 (pmol/L). GLP-1 concentration in serum will be determined in duplicate via enzyme-linked immunosorbent assay kits (ELISA; Millipore, Billerica, Massachusetts).

CONTACTS AND LOCATIONS:
Overall Officials: Nick Bellissimo, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- School of Nutrition, Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided